CLINICAL TRIAL: NCT06955949
Title: Comparison Of Mobilization With Movement And ESWT Treatment Modalities In Patients With Lateral Epicondylopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LE-MWM-ESWT-2025-01
Record Dates: First submitted 2025-04-15; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Effects of MWM and ESWT on Pain and Function in LE Patients
Keywords: Lateral Epicondylopathy; ESWT; Mobilization with Movement
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Active Comparator): Eccentric strengthening exercises (3 sets of 10 repetitions) with dumbbells were performed as distributed in the control groups.
  Interventions: Other: Control Group
- ESWT group (Active Comparator): ESWT group will receive Extracorporeal Shock Wave Therapy, a noninvasive treatment that uses acoustic waves to promote healing and reduce pain in musculoskeletal disorders
  Interventions: Other: ESWT Group
- MWM (Active Comparator): Mobilization with Movement Technique Group "MWM is a manual therapy technique that includes active movement combined with mobilization applied by the therapist to reduce fragmentation and pain.
  Interventions: Other: Mobilization movement group
- Combined MWM-ESWT group (Active Comparator): Mobilization with Movement and ESWT Group The combined MWM + ESWT group will receive Mobilization with Movement (MWM), a manual therapy technique for comprehensive function and pain reduction, and Extracorporeal Shock Wave Therapy (ESWT), a noninvasive treatment that uses acoustic waves to promote healing and reduce musculoskeletal pain.
  Interventions: Other: Combined MWM-ESWT

INTERVENTIONS:
Other: Control Group — The control classes applied the drugs by doing home training with eccentric strengthening exercises with dumbbells (3 sets of 10 repetitions). They were asked to flex the wrist while the wrist was fully extended. Weights were given to strengthen the wrist extensor muscles with 0.5 kg in the first week, 1 kg in the second week and 1.5 kg in the third week. In addition, stretching exercises for the wrist extensor muscles (3 sets of 20 seconds) were performed and 20 seconds of rest were given between sets. After the exercises, we applied cold therapy for 15 minutes. All treatment types were treated by the same physiotherapist in accordance with the treatment protocols and treatment sessions were performed twice a week for 3 weeks. One session lasted between 35-45 minutes.
  Arms: Control group
Other: ESWT Group — Extracorporeal Shock Wave Therapy (ESWT) is palpated at the starting areas of the extensor carpi radialis brevis and longus muscles, at tender points, and placed at the bone-tendon junctions. This budget was set at 90 Hz, and the pulse rate was determined as 10 pulses:1500.
  Arms: ESWT group
Other: Mobilization movement group — Mobilization Technique (lateral glide) was recorded from the Mulligan method. Patients were placed in supine positions, height was recorded together and the application was done with a belt method. During this glide movement, the patient was asked to actively perform 3 sets of 10 repetitions of wrist extension. 15-20 seconds of rest was given between sets.
  Arms: MWM
Other: Combined MWM-ESWT — In addition to mobilization with movement and ESWT treatment, this group applied home training by doing eccentric exercises with dumbbells (3 sets of 10 repetitions). 15-20 seconds of rest was given between sets. In addition, stretching exercises (3 sets of 20 seconds) were performed to strengthen the wrist extensor muscles and 20 seconds of rest was given between sets. During the exercises, a position was given such that the elbow was in extension, the forearm was in pronation and the wrist was in ulnar deviation. We apply cold therapy for 15 minutes after the exercises.
  Arms: Combined MWM-ESWT group

SUMMARY:
Abstract Our study aimed to compare the effects of mobilization with movement (MWM) and extracorporeal shock wave therapy (ESWT) on pain and functionality in patients with lateral epicondylopathy. A total of 57 volunteers aged 18-65 years, diagnosed with lateral epicondylopathy and referred to the clinic, were divided into groups. In the mobilization with movement group, patients performed active wrist extension exercises using a dumbbell (3 sets of 10 repetitions) while lateral glide mobilization was maintained. In the ESWT group, the therapy was administered at a frequency of 90 Hz and a pulse rate of 10 pulses per 1500. A separate group received a combination of mobilization with movement and ESWT. Additionally, strengthening and stretching exercises, along with cold pack application (15 minutes), were provided twice a week for three weeks to all groups, including the control group. Pain intensity was assessed using the Visual Analog Scale (VAS), and functionality was evaluated using the PRTEE-T (Patient Rated Tennis Elbow Evaluation- Turkish Version ) questionnaire. The Upper Extremity Y-Balance Test was also performed before and after treatment, and all measurements were recorded.

The findings of our study revealed that, in between-group comparisons, the mobilization with movement group demonstrated superior outcomes in pain reduction (resting and nighttime), PRTEE, and Upper Extremity Y-Balance Test performance compared to other groups.

Keywords: Lateral Epicondylopathy, ESWT, Mobilization with Movement

DETAILED DESCRIPTION:
Introduction Lateral epicondylopathy was first described by Dr. Runge in 1873 as "tennis elbow" . Although previously referred to as "lateral epicondylitis" in earlier research, recent studies have updated the term to "lateral epicondylopathy" .

The exact cause of lateral epicondylopathy remains unclear, but it is thought to result from overuse of the forearm extensor muscles, leading to microtears in the extensor carpi radialis brevis tendon or direct trauma .

Difficulties experienced during daily activities are among the most common complaints of patients. The diagnosis of lateral epicondylopathy can be easily made through specific tests and a detailed patient history. Severe pain during resisted wrist extension, third finger extension, and passive wrist flexion, as well as movement restriction, tenderness at the lateral epicondyle, and reduced grip strength, are among the findings supporting the diagnosis .

The primary goal of treating lateral epicondylopathy is to reduce the patient's current pain and enable them to return to daily activities as soon as possible. Conservative treatment methods achieve a 95% success rate. These approaches include rest, non-steroidal anti-inflammatory drugs (NSAIDs), corticosteroid injections, intermittent ultrasound (US), transcutaneous electrical nerve stimulation (TENS), orthotic devices, myofascial release techniques, transverse friction massage, mobilization, kinesiology taping (KT), cold application, and extracorporeal shock wave therapy (ESWT) Treatments for lateral epicondylopathy are generally classified as either surgical or non-surgical.

One of the conservative treatment methods, ESWT, has been used for years in the treatment of orthopedic disorders. The primary goal of this method is to enhance circulation and activate healing mechanisms by focusing high-intensity sound waves on the target area . Although many studies in the literature support the efficacy of ESWT, some randomized controlled trials have suggested that this treatment may be ineffective or no different from a placebo effect. For example, in a study by Bryan Chung et al., ESWT was compared with forearm stretching exercises, and no significant difference was found between the two methods .

The Mobilization with Movement (MWM) technique is an innovative manual therapy method developed by Mulligan. This technique is widely preferred for correcting improper elbow positioning. Unlike traditional treatments, this method involves lateral gliding mobilization while ensuring pain-free grip and wrist extension, ultimately improving elbow functionality. The Mulligan technique can be safely applied to the musculoskeletal and nervous systems, integrating multiple treatment approaches. Its main advantage is that it provides both short-term and long-term functional mobility improvements.

This study aims to compare the effectiveness of the MWM technique and ESWT in patients with lateral epicondylopathy and to evaluate the effects of these methods on pain, movement restriction, and functionality.

Methods Participants and Study Design This study aimed to compare the effects of the mobilization with movement (MWM) technique and extracorporeal shock wave therapy (ESWT) treatment modalities on pain, movement restriction, and functionality in patients with lateral epicondylopathy. The research included 57 voluntary patients aged 18-65 who were diagnosed with lateral epicondylopathy and admitted to the Physical Therapy Clinic of Yalova Çınarcık State Hospital.

The inclusion criteria included complaints persisting for at least three months, tenderness in the lateral epicondyle region, decreased strength in the extensor carpi radialis brevis (ECRB) muscle, increased pain during resisted wrist extension, pain on the lateral side of the elbow, and discomfort triggered by repetitive rotational movements. The exclusion criteria included the presence of multiple elbow problems, previous elbow joint surgery, tendon rupture, joint movement restriction due to humerus, radius, or ulna fractures, cervical radiculopathy, difficulty in cooperation, or refusal to participate in the study.

Ethical approval was obtained from the İstinye University Clinical Research Ethics Committee (3/2022.K-09), and written informed consent forms were collected from all participants. The study was designed as a randomized parallel-controlled experimental trial. Sample size calculation was performed using G-Power analysis, targeting 56 participants with 80% power, a 5% type 1 error rate, and a moderate effect size (0.40). A total of 60 individuals meeting the criteria were initially included, but three participants were unable to complete the final assessment due to personal reasons. The study was ultimately completed with 57 individuals.

Participants were divided into four groups, each consisting of 15 individuals:

* Mobilization with Movement (MWM) group
* ESWT group
* Combined MWM + ESWT group
* Control group Evaluation and Test Protocols

  1. Pain Assessment Pain assessment was conducted using the Visual Analog Scale (VAS), a widely used technique for measuring pain intensity. Patients marked their pain levels on a 10 cm-long line, where 0 represented no pain, and 100 represented maximum pain .
  2. PRTEE (Patient-Rated Tennis Elbow Evaluation) Questionnaire for Functional Assessment The PRTEE questionnaire was used to assess functional levels in patients with lateral epicondylopathy. This questionnaire consists of two main sections evaluating pain and functional limitations in the affected arm. Pain and function scores range from 0-50 each, with a total score ranging from 0 to 100, where higher values indicate worse conditions.
  3. Upper Extremity Y-Balance Test The Y-Balance Test was used to assess dynamic balance. The test involves reaching movements in three directions (medial, inferolateral, and superolateral). Participants assumed a push-up position and attempted to reach designated points with the tested hand. The reached distances were recorded in centimeters, and the composite score was calculated as follows: Composite Score = (Medial + Inferolateral + Superolateral Reach Distance) / Arm Length × 100 .

Treatment Protocols

All patients participating in the study were informed about the movements they should avoid during the treatment period. These movements include wringing clothes, prolonged computer use, gardening, and heavy lifting.

Mobilization with Movement Technique Group

The mobilization technique (lateral glide) from the Mulligan method was used. Patients were placed in a supine position, in a pain-free position, and the application was performed with the assistance of a belt. During this glide movement, the patient was asked to actively perform 3 sets of 10 repetitions of wrist extension. Rest periods of 15-20 seconds were given between sets.

ESWT Group

Extracorporeal Shock Wave Therapy (ESWT) was applied at the bone-tendon junctions of the extensor carpi radialis brevis and longus muscles' origin areas, where sensitive points were palpated. In this application, the frequency was set to 90 Hz, and the pulse rate was set to 10 pulses:1500.

Mobilization with Movement and ESWT Group

This group, in addition to mobilization with movement and ESWT treatment, performed eccentric strengthening exercises with dumbbells (3 sets of 10 repetitions) as homework. Rest periods of 15-20 seconds were given between sets. Additionally, stretching exercises (3 sets of 20 seconds) were performed to strengthen the wrist extensor muscles, with rest periods of 20 seconds between sets. During exercises, a position was given where the elbow was extended, the forearm was pronated, and the wrist was in ulnar deviation. After the exercises, 15 minutes of cold therapy was applied.

Control Group

Patients in the control group performed eccentric strengthening exercises with dumbbells (3 sets of 10 repetitions) as homework. While the wrist was in full extension, they were asked to perform wrist flexion with 0.5 kg in the first week, 1 kg in the second week, and 1.5 kg in the third week, to strengthen the wrist extensor muscles. Additionally, stretching exercises (wrist extensors) were performed for 3 sets of 20 seconds, with 20-second rest periods between sets. After the exercises, 15 minutes of cold therapy was applied.

All treatment groups were treated by the same physiotherapist according to the treatment protocols, with treatment sessions twice a week for 3 weeks. Each session lasted between 35-45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Continuation of complaints for at least 3 months
* Tenderness over the lateral epicondyle
* Decreased ECRB muscle strength
* İncreased pain during resisted extension of the wrist
* Pain complaints on the lateral side of the elbow
* Pain resulting from repetitive and especially rotational movements

Exclusion Criteria:

* Having a different elbow problem or more than one elbow problem
* Having had elbow joint surgery
* Having tendon rupture
* Having a history of humerus
* Radius or ulna fractures
* Having limited range of motion known
* Having cervical radiculopathy
* Having difficulty in cooperation and refusing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity, assessed by the Visual Analog Scale (VAS) Because pain reduction (resting and nighttime) is the most emphasized and statistically analyzed main outcome in the study, it is considered the primary outcome. | Baseline (Pre-treatment) and Week 3 (Post-treatment)
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a 10 cm line on which participants mark their perceived pain level, ranging from "no pain" (0) to "worst imaginable pain" (10). Both resting pain and nighttime pain will be evaluated.

SECONDARY OUTCOMES:
Functional Status (PRTEE-T) | Baseline (Pre-treatment) and Week 3 (Post-treatment)
  Functionality will be evaluated using the Patient-Rated Tennis Elbow Evaluation - Turkish version (PRTEE-T) questionnaire. This tool assesses pain and functional limitations associated with lateral epicondylopathy. Scores range from 0 to 100, with higher scores indicating greater disability.
Upper Extremity Performance (Y-Balance Test) | Baseline (Pre-treatment) and Week 3 (Post-treatment)
  Upper extremity performance will be assessed using the Upper Extremity Y-Balance Test. Participants reach in three directions (medial, inferolateral, superolateral) while in a push-up position. Reach distances are measured in centimeters and used to calculate a composite score that reflects dynamic balance and functional performance

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol